CLINICAL TRIAL: NCT05619302
Title: Molecular Imaging of Myocardial Fibrosis in Cardiac Amyloidosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sharmila Dorbala, Director of Nuclear Cardiology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022A012856
Record Dates: First submitted 2022-11-09; First posted 2022-11-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Amyloidosis
Keywords: Amyloidosis; Cardiac; Heart; Imaging; Diagnosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- [68Ga]CBP8 PET/MRI Amyloid Subjects (Experimental): Individuals with documented cardiac amyloidosis will undergo [68Ga]CBP8 PET/MRI.
  Interventions: Drug: [68Ga]CBP8 PET/MRI
- [68Ga]CBP8 PET/MRI Recent Myocardial Infarction Subjects (Active Comparator): Individuals with recent myocardial infarction will undergo [68Ga]CBP8 PET/MRI.
  Interventions: Drug: [68Ga]CBP8 PET/MRI
- [68Ga]CBP8 PET/MRI Healthy Controls (Placebo Comparator): Individuals without documented cardiovascular disease will undergo [68Ga]CBP8 PET/MRI.
  Interventions: Drug: [68Ga]CBP8 PET/MRI
- [68Ga]CBP8 PET/MRI Hypertrophic Cardiomyopathy Subjects (Active Comparator): Individuals with hypertrophic cardiomyopathy will undergo [68Ga]CBP8 PET/MRI.
  Interventions: Drug: [68Ga]CBP8 PET/MRI

INTERVENTIONS:
Drug: [68Ga]CBP8 PET/MRI — Simultaneous cardiac PET/MRI images will be obtained following injection of [68Ga]CBP8
  Other Names: No other names

SUMMARY:
The primary aim of our pilot study is to determine whether fibrosis in the heart can be measured with [68Ga]CBP8, a positron emission tomography (PET) probe, using PET/magnetic resonance imaging (MRI) imaging, in 30 individuals with documented cardiac amyloidosis. The investigators will also enroll 15 individuals with recent myocardial infarction and 15 individuals with hypertrophic cardiomyopathy as positive controls for fibrosis, and the investigators will enroll 5 individuals without cardiovascular disease to undergo [68Ga]CBP8 PET/MRI imaging as a healthy control group.

The primary hypothesis of this study is that [68Ga]CBP8 will bind to interstitial collagen and quantify myocardial fibrosis in patients with cardiac amyloidosis. The investigators hypothesize that [68Ga]CBP8 uptake will be greater in patients with cardiac amyloidosis, myocardial fibrosis, and hypertrophic cardiomyopathy than in healthy controls. Secondly, the investigators also hypothesize that [68Ga]CBP8 activity more strongly correlates with standard MRI measures in patients with recent myocardial infarction and hypertrophic cardiomyopathy (where extracellular expansion is caused by myocardial fibrosis/collagen deposition) than in patients with cardiac amyloidosis (where myocardial fibrosis is combined with infiltration).

DETAILED DESCRIPTION:
[68Ga]CBP8 is a novel gallium-68 labeled positron emission tomography (PET) probe that selectively binds collagen type I, which constitutes the majority of fibrotic tissue. In pre-clinical mouse models, [68Ga]CBP8 had the sensitivity to detect pulmonary fibrosis even at early stages and specificity for collagen uptake with low non-specific uptake in background tissues and organs. In preliminary studies in humans with idiopathic pulmonary fibrosis, patients tolerated [68Ga]CBP8 without adverse effects, and there was a strong correspondence between high collagen tracer signal and fibrotic lung regions established by chest computed tomography (CT) scan. [68Ga]CBP8 may be a valuable tool to detect and quantify collagen in the heart. The investigators propose to test [68Ga]CBP8 in a pilot study to image myocardial fibrosis in patients with cardiac amyloidosis.

Cardiac amyloidosis is characterized by myocardial interstitial infiltration by misfolded amyloid fibrils. Infiltration leads to increased myocardial stiffness and heart failure. In patients with cardiac amyloidosis, myocardial stiffness may also be caused by extracellular collagen deposition in the myocardium. Collagen deposition (i.e. myocardial fibrosis) results in adverse cardiac remodeling through similar mechanisms as amyloidosis and may potentiate heart failure in patients with cardiac amyloidosis. Myocardial fibrosis can be mitigated or prevented. In addition, therapies directed against amyloid fibrils also have differential response rates in cardiac amyloidosis patients with or without coexistent fibrosis. Magnetic resonance imaging (MRI) is an established method of measuring extracellular volume (ECV), a reliable way of quantifying myocardial fibrosis in conditions where the primary reason for ECV expansion is myocardial fibrosis. ECV may not be an optimal surrogate of myocardial fibrosis in patients with cardiac amyloidosis, where ECV is already quite expanded due to myocardial amyloid infiltration. Thus, a means of accurate, non-invasive quantitation of myocardial fibrosis has the potential to significantly improve cardiac amyloidosis care.

This pilot study is designed to understand whether myocardial fibrosis can be measured using a collagen 1 targeted radiotracer ([68Ga]CBP8). The investigators would like to study 15 patients with light-chain (AL) cardiac amyloidosis and 15 patients with transthyretin (ATTR) cardiac amyloidosis to understand differences in radiotracer uptake, if any. The investigators will also enroll 15 patients with recent myocardial infarction and 15 patients with hypertrophic cardiomyopathy as positive controls for fibrosis and will enroll 5 individuals without cardiovascular disease as negative controls.

The aim of this proposed research study is, using simultaneous PET/MRI imaging, to determine whether [68Ga]CBP8 uptake will accurately identify and quantify myocardial fibrosis in patients with cardiac amyloidosis, recent myocardial infarction, and hypertrophic cardiomyopathy. The aim of this study is also to correlate [68Ga]CBP8 PET uptake with standard MRI measures in patients with cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria for AL-amyloid subjects:

* Age > 18 years
* Willing and able to provide consent
* AL-CA: Diagnosis of systemic light chain amyloidosis by standard criteria: Immunofixation of serum, serum free light chain (FLC) assay, a biopsy of fat pad/bone marrow, or organ biopsy, followed by typing of the light chain using immunohistochemistry or immunogold assay with confirmation by mass spectroscopy as needed AND

  * Proof of cardiac involvement by AL amyloidosis
  * Abnormal cardiac biomarkers: abnormal high sensitivity TnT 5th generation levels (> 15 ng/L) or abnormal age-appropriate NT-proBNP (abnormal values: < 50 years: > 450 pg/ml; 50-75 years: > 900 pg/ml; > 75 years: > 1800 pg/ml) OR
  * Abnormal echocardiogram (wall thickness > 12 mm in the absence of other causes of increased LV wall thickness) OR
  * Abnormal CMR (wall thickness > 12 mm, extracellular volume > 0.40 or typical CMR appearance of cardiac amyloidosis with difficulty nulling images and non-coronary distribution late gadolinium enhancement) OR
  * Positive endomyocardial biopsy

Inclusion Criteria for ATTR-amyloid subjects:

* Age > 18 years
* Willing and able to provide consent
* ATTR-CA: Diagnosis of either wildtype or hereditary transthyretin cardiac amyloidosis by standard criteria: Endomyocardial biopsy followed by typing of the transthyretin amyloidosis using immunohistochemistry or immunogold assay with confirmation by mass spectroscopy as needed

  * Extracardiac biopsy with typical cardiac imaging findings
  * Hereditary ATTR amyloidosis by genetic testing OR
  * Grade 2 or grade 3 myocardial uptake of 99mTc-PYP if AL amyloidosis is excluded

Inclusion Criteria for recent myocardial infarction subjects:

* Age > 18 years
* Willing and able to provide consent
* Recent MI: Diagnosis of recent type 1 myocardial infarction by standard criteria

  * More than 6 weeks from diagnosis of MI but within 6 months
  * Imaging evidence of loss of viable myocardium or persistent regional wall motion abnormalities in a pattern consistent with an ischemic etiology in more than one segment

Inclusion Criteria for hypertrophic cardiomyopathy subjects:

* Age > 18 years
* Willing and able to provide consent
* Hypertrophic cardiomyopathy: Diagnosis of hypertrophic cardiomyopathy by standard criteria
* MRI evidence of late gadolinium enhancement

Inclusion Criteria for recent healthy control subjects:

* Age > 18 years
* Willing and able to provide consent
* No known cardiac amyloidosis or recent myocardial infarction

Exclusion Criteria:

* Dialysis
* NYHA (New York Heart Association) Class IV
* Acute myocardial infarction within 6 weeks
* Pregnancy or nursing
* History of adverse events from or allergy to gadolinium contrast media
* Hemodynamic instability
* Severe claustrophobia despite use of sedatives
* Decompensated heart failure (unable to lie flat for 1 hour)
* Concomitant clinically significant non-ischemic non-amyloid heart disease (valvular heart disease or dilated cardiomyopathy)
* Body weight over limit for MRI table (>300 lbs)
* Contraindications for MRI (including non-compatible cardiac implantable electronic devices, drug infusion pumps, and metallic or electric implants)
* Any other reason determined by the investigator to be unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Standardized Uptake Value (SUVmean) of [68Ga]CBP8 uptake in the heart | 1 day
  Standardized uptake value (SUV) mean is defined as the mean [68Ga]CBP8 concentration measured within the left ventricular myocardium multiplied by the decay-corrected amount of injected [68Ga]CBP8 normalized to patient weight. We expect SUVmean will be greater in patients with cardiac amyloidosis and myocardial infarction compared with healthy control subjects.
Extracellular volume from clinically performed simultaneous cardiac MRI | 1 day
  We will correlate [68Ga]CBP8 uptake with standard MRI extracellular volume (ECV) measures. We expect [68Ga]CBP8 activity to more strongly correlate with MRI in patients with myocardial infarction than cardiac amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Dorbala, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Desogere P, Tapias LF, Rietz TA, Rotile N, Blasi F, Day H, Elliott J, Fuchs BC, Lanuti M, Caravan P. Optimization of a Collagen-Targeted PET Probe for Molecular Imaging of Pulmonary Fibrosis. J Nucl Med. 2017 Dec;58(12):1991-1996. doi: 10.2967/jnumed.117.193532. Epub 2017 Jun 13. PMID 28611243
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537